CLINICAL TRIAL: NCT06725511
Title: Wellness Program Outreach and Effectiveness: A Randomized Controlled Trial
Brief Title: Wellness Program Outreach and Effectiveness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other); Quest Diagnostics-Nichols Insitute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2402001204
Record Dates: First submitted 2024-11-22; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Workplace wellness
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opt-in Outreach (Active Comparator): Outreach notifies those eligible that they are invited to join the program, as usual practice.
  Interventions: Behavioral: Opt-in framing
- Opt-out Outreach (Experimental): Outreach notifies those eligible that they are enrolled in the program and invited to begin their first session.
  Interventions: Behavioral: Opt-out framing

INTERVENTIONS:
Behavioral: Opt-out framing — Outreach notifies those eligible that they are enrolled in the program and invites them to start participating.
  Arms: Opt-out Outreach
Behavioral: Opt-in framing — Eligible participants are invited to enroll
  Arms: Opt-in Outreach

SUMMARY:
The investigators will conduct a randomized controlled trial to evaluate the impact of an outreach campaign designed to increase engagement with Pack Health, a Quest Diagnostics wellness program providing individual health coaching for weight management and diabetes prevention. While employee wellness and disease-management programs have the potential to improve wellbeing and reduce healthcare costs, their effectiveness is often undermined by low engagement and selection bias in participant comparisons. This study will test whether an outreach approach that auto-enrolls eligible individuals-employees and their spouses/domestic partners-into the program, with the option to opt out, can increase engagement and improve health outcomes compared to the standard invitation-based approach.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial to evaluate the impact of an outreach campaign designed to increase engagement with Pack Health, a Quest Diagnostics wellness program providing individual health coaching for weight management and diabetes prevention. While employee wellness and disease-management programs have the potential to improve wellbeing and reduce healthcare costs, their effectiveness is often undermined by low engagement and selection bias in participant comparisons. This study will test whether an outreach approach that auto-enrolls eligible individuals-employees and their spouses/domestic partners-into the program, with the option to opt out, can increase engagement and improve health outcomes compared to the standard invitation-based approach.

Participants will be randomly assigned to one of two groups: the intervention group, which will receive auto-enrollment outreach, and the control group, which will receive traditional invitation-based outreach. The primary outcome will measure program engagement as the share who begin the program. Secondary outcomes will include additional measures of engagement, such as the number of modules completed, health outcomes observed in subsequent risk assessments and healthcare claims, and employee retention. This trial will provide evidence on whether an opt-out framing in outreach campaigns can enhance the effectiveness of wellness programs, ultimately informing best practices for population health management.

ELIGIBILITY:
Inclusion Criteria:

1. Provided informed consent.
2. Those who are eligible for the Pack Health program:

   * Employees/spouses/domestic partners over the age of 18
   * Metabolic syndrome defined as results indicating 3 or more of the following risk factors:

     * High waist circumference (>35 inches for women and >40 inches for men)
     * High triglycerides (≥150 mg/dl)
     * Low HDL cholesterol (<50 mg/dl for women and <40 mg/dl for men)
     * High Blood Pressure (≥130/85)
     * High Fasting Glucose (≥100 mg/dl)

Exclusion Criteria:

* 1. Anyone under the age of 21. They will not be part of the study and will receive messages as if they were in the control group.

  2. Anyone observed in claims data with a historical diagnosis of:
  * Anorexia nervosa
  * Bulimia nervosa
  * Binge-eating disorder
  * Body dysmorphic disorder
  * Major depression
  * Post-traumatic stress disorder (PTSD)
  * Severe anxiety disorder

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Probability of Engagement initiation | 12 months
  The outcome is whether participants begin the program at some point during the Annual Risk Assessment year.

SECONDARY OUTCOMES:
Probability of Engagement level | 12 months
  Number of modules completed during the Annual Risk Assessment year.
Probability of Retention at end of annual-risk-assessment year | 12 months
  Indicator the person is working for the firm on August 31, 2025
Annual Risk Assessment Measures: HbA1c | 24 months
  HbA1c the following year's Annual Risk Assessment
Annual Risk Assessment Measures: Weight | 24 months
  Weight measured in the following year's Annual Risk Assessment

OTHER OUTCOMES:
Probability of full program engagement | 12 months
  Indicator for completing 9 modules during the Annual Risk Assessment year.
Probability of membership in the top 5% of healthcare claims | 12 months
  Indicator that the person is in the right tail of the distribution of claims.
Probability of membership in the top 1% of healthcare claims | 12 months
  Indicator that the person is in the right tail of the distribution of claims.
Mean number of Inpatient visits | 12 months
  Number of inpatient visits during the Annual Risk Assessment year.
Mean number of ED visits | 12 months
  Number of emergency department visits during the Annual Risk Assessment year.
Mean number of outpatient visits | 12 months
  Number of outpatient visits during the Annual Risk Assessment year.
Mean total healthcare claims | 12 months
  Total healthcare claims during the Annual Risk Assessment year.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Doyle, PhD, Principal Investigator — MIT Sloan School of Management
Locations (1):
- Quest Diagnostics, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Subject to approval from implementation partner.

DOCUMENTS (2):
  • Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT06725511/SAP_000.pdf
  • Informed Consent Form (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT06725511/ICF_001.pdf